CLINICAL TRIAL: NCT04977167
Title: A Phase I Open Label Study of HG146 Alone /in Combination with PD-(L)1 Inhibitor Administered with and Without Anticancer Agents in Participants with Advanced Solid Tumors or Lymphoma
Brief Title: Clinical Trial of HG146 Administered to Subjects with Advanced Solid Tumors or Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HitGen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HG146CN102
Record Dates: First submitted 2021-07-12; First posted 2021-07-26 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1:HG146 Monotherapy, Dose-escalation Cohort (Experimental): Subjects will receive HG146 PO at every two days intervals (qod) for 14 consecutive days,7 days off, 21 days/ cycle. Escalating doses of HG146 will be evaluated using 3+3 approach.
  Interventions: Drug: HG146
- Part 2A:HG146 + PD-(L)1 antibody, Dose escalation Cohort (Experimental): Subjects will receive HG146 PO at every two days intervals (qod) for 14 consecutive days,7 days off, along with PD-(L)1 antibody IV once every 3 weeks (Q3W),21 days/ cycle.
  Escalating doses of HG146 in combination with PD-(L)1 antibody will be evaluated.
  Interventions: Drug: HG146; Drug: PD-(L)1 antibody
- Part 2B-1：HG146 combination Expansion Cohort 1 (Experimental): Subjects who have not been treated with PD-(L)1 antibody，will receive HG146 po for 14 consecutive days,7 days off, in combination with PD-(L)1 antibody IV Q3W.
  Interventions: Drug: HG146; Drug: PD-(L)1 antibody
- Part 2B-2：HG146 combination Expansion Cohort 2 (Experimental): Subjects who have progressed on PD-(L)1 antibody, will receive HG146 po for 14 consecutive days,7 days off, in combination with PD-(L)1 antibody IV Q3W.
  Interventions: Drug: HG146; Drug: PD-(L)1 antibody

INTERVENTIONS:
Drug: HG146 — HG146 is available as Capsule at a unit dose strength of 5 mg and 10 mg.
Drug: PD-(L)1 antibody — PD-(L)1 Antibody is available as solution for infusion or lyophilized powder for reconstitution to be administered Q3W. It will be administered as an IV infusion for 30 minutes.
  Arms: Part 2A:HG146 + PD-(L)1 antibody, Dose escalation Cohort; Part 2B-1：HG146 combination Expansion Cohort 1; Part 2B-2：HG146 combination Expansion Cohort 2

SUMMARY:
This is a Phase I, open-label, repeat-dose, non-randomized, multicenter study to evaluate the safety, tolerability, and preliminary clinical activity and establish a recommended dose of HG146 administered orally (PO) alone (Part 1) or co-administered (Part 2) with PD-（L）1 inhibitor in subjects with refractory/relapsed solid tumors or Lymphoma. Part 1 consists of a dose escalation phae,Part2 consists of a dose escalation phase and a cohort expansion phase. In Part 1, escalating doses of HG146 will be evaluated as guided by the "3+3" approach. In Part 2A, escalating doses of HG146 in combination with PD-(L)1 inhibitor will be evaluated as guided by the "3+3" approach. In Part 2B, subjects will receive a single dose level of HG146 as identified based on data from Part 2, in combination with PD-(L)1 inhibitor . A total of approximately 96 subjects will be enrolled in this study, approximately 36 for dose escalation cohorts, and approximately 60 in the expansion cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

1 Subject must be >=18 years of age at the time of signing the informed consent.

2- Ia/Ib dose escalation phase（Part1 and Part 2A）：Subjects with advanced/Metastatic solid tumors or Lymphoma, who have progressed on, be intolerant of, or ineligible for, all available therapies for which clinical benefit has been established.

* Ib dose expansion phase（Part 2）:

  1. Cohort 1,Subjects with advanced/Metastatic solid tumors or Lymphoma, who have progressed on, be intolerant of, or ineligible for, all available therapies for which clinical benefit has been established, have not been treated with PD-(L)1 antibody； 2）Cohort 2,Subjects with advanced/Metastatic solid tumors or Lymphoma, who have progressed on, be intolerant of, or ineligible for, all available therapies for which clinical benefit has been established, have progressed on PD-(L)1 antibody； 3 Measurable disease per RECIST version 1.1 or Lugano 2014（If applicable）. 4 Has Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1. 5 Has adequate organ function. 6 Signed informed consent form (ICF) and able to comply with study requirements.

Key Exclusion Criteria:

1. Received prior therapies targeting HDAC.
2. Symptomatic central nervous system (CNS) metastases that have required steroids within 4 weeks prior to first dose of study treatment.
3. History of intolerant of anti-PD-(L)1 toxicity（Ib）.
4. A condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of enrollment.
5. Major surgery or major injury <=28 days before the first dose of study treatment,or anticipated major surgery during the study.
6. Received other anticaner therapies within 4 weeks prior to first dose of study treatment or 5 half life period of anticancer drug .
7. Active infection requiring systemic treatment.
8. Prior allogeneic bone marrow transplantation or other solid organ transplantation ( Ib)
9. Active autoimmune disease or disease of impaired immune system(Ib).
10. History of Adrenal insufficiency.(Ib)
11. History orConcurrent condition of other malignant tumors.
12. Recent (within the past 6 months) history of Unstable or serious diseases, such as pancreatitis, severe angina, prolonged QT interval, congestive heart failure, myocardial infarction, pulmonary hypertension, stroke, and severe seizures, etc.
13. History of severe lung disease.
14. Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his/her compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Part 1:Number of participants experiencing Dose-Limiting Toxicities (DLTs) According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v.5.0) | Up to 26 Days in Cycle 0 and Cycle 1
Part 1:Number of participants experiencing Serious Adverse Events (SAEs) and Adverse Events (AE) | Up to 2 years
Part1:Maximum tolerated dose or Recommended Phase Ib dose (RP2D) of HG146 | Up to 2 years
Part 2A:Number of participants experiencing Dose-Limiting Toxicities (DLTs) According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v.5.0) | Up to 21 Days in Cycle 1
Part 2A:Number of participants experiencing Serious Adverse Events (SAEs) and Adverse Events (AE) | Up to 2 years
Part 2A:Maximum tolerated dose or Recommended Phase Ib dose (RP2D) of HG146 in combination with PD-(L)1 antibody | Up to 2 years

SECONDARY OUTCOMES:
Part 1:Area under the concentration versus time curve (AUC) of HG146 | At the end of Cycle 0 Day 5 (Cycle 0 is 5 days);At the end of Cycle 1 Day15 (Except for cycle 0, each cycle is 21 days)
  Plasma concentration of HG146 will be measured following single dose and multiple dose administration
Part 1:Peak plasma concentration (Cmax) of HG146 | At the end of Cycle 0 Day 5 (Cycle 0 is 5 days);At the end of Cycle 1 Day15 (Except for cycle 0, each cycle is 21 days)
  Plasma concentration of HG146 will be measured following single dose and multiple dose administration
Part 1:Time of Cmax (Tmax) of HG146 | At the end of Cycle 0 Day 5 (Cycle 0 is 5 days);At the end of Cycle 1 Day15(Except for cycle 0, each cycle is 21 days)
  Plasma concentration of HG146 will be measured following single dose and multiple dose administration
Part 1:Apparent terminal half-life (T1/2) of HG146 | At the end of Cycle 0 Day 5 (Cycle 0 is 5 days);At the end of Cycle 1 Day15 (Except for cycle 0, each cycle is 21 days)
  Plasma concentration of HG146 will be measured following single dose and multiple dose administration
Part1: objective response rate (ORR) | Up to 2 years
  ORR will be assessed by the Investigators using RECIST v. 1.1 or Lugano 2014( If applicable)
Part1: Best overall response (BOR) | Up to 2 years
  BOR will be assessed by the Investigators using RECIST v. 1.1 or Lugano 2014( If applicable)
Part1: Duration of response (DOR) | Up to 2 years
  DOR will be assessed by the Investigators using RECIST v. 1.1 or Lugano 2014( If applicable)
Part 1:Time-to-response (TTR) | Up to 2 years
  TTR will be assessed by the Investigators using RECIST v. 1.1 or Lugano 2014( If applicable)
Part 1:Progression-Free Survival (PFS) | Up to 2 years
  PFS will be assessed by the Investigators using RECIST v. 1.1 or Lugano 2014( If applicable)
Part 2:Area under the concentration versus time curve (AUC) of HG146 | At the end of Cycle 1 Day 15 (each cycle is 21 days)
  Plasma concentration of HG146 will be measured following multiple dose administration in combination with PD-(L)1 antibody
Part 2:maximum observed plasma concentration (Cmax) of HG146 | At the end of Cycle 1 Day 15 (each cycle is 21 days)
  Plasma concentration of HG146 will be measured following multiple dose administration in combination with PD-(L)1 antibody
Part 2:time of maximum observed plasma concentration (Tmax) of HG146 | At the end of Cycle 1 Day 15 (each cycle is 21 days)
  Plasma concentration of HG146 will be measured following multiple dose administration in combination with PD-(L)1 antibody
Part 2:apparent terminal half-life (T1/2) of HG146 | At the end of Cycle 1 Day 15 (each cycle is 21 days)
  Plasma concentration of HG146 will be measured following multiple dose administration in combination with PD-(L)1 antibody
Part2: objective response rate (ORR) | Up to 2 years
  ORR will be assessed by the Investigators using RECIST v. 1.1 or Lugano 2014( If applicable)
Part2: Best overall response (BOR) | Up to 2 years
  BOR will be assessed by the Investigators using RECIST v. 1.1 or Lugano 2014( If applicable)
Part2: Duration of response (DOR) | Up to 2 years
  DOR will be assessed by the Investigators using RECIST v. 1.1 or Lugano 2014( If applicable)
Part 2:Time-to-response (TTR) | Up to 2 years
  TTR will be assessed by the Investigators using RECIST v. 1.1 or Lugano 2014( If applicable)
Part 2:Progression-Free Survival (PFS) | Up to 2 years
  PFS will be assessed by the Investigators using RECIST v. 1.1 or Lugano 2014( If applicable)
OS | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — National Cancer Center/Cancer Hospital
Locations (1):
- National Cancer Center/Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No